CLINICAL TRIAL: NCT06499272
Title: Quality-of-Life-and-Cognitive-Oriented Rehabilitation Program Through the NeuronUP in Older People With Alzheimer's Disease: A Randomized Clinical Trial
Brief Title: Quality-of-Life-and-Cognitive-Oriented Rehabilitation Through the NeuronUP in Alzheimer's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Rey Juan Carlos (Other)
Responsible Party: Principal Investigator, Cristina García-Bravo, PhD, Occupational Therapist, Universidad Rey Juan Carlos
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 271120234112023
Record Dates: First submitted 2024-07-06; First posted 2024-07-12 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-07

CONDITIONS: Alzheimer Disease; Occupational Therapy; Quality of Life; Cognitive Impairment; Older People
Keywords: Alzheimer's Disease; Occupational Therapy; NeuronUP; Quality of Life; Cognitive Stimulation; Cognitive Impairment
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: ontrol Group (CG), which received their usual sessions of conventional occupational therapy, and an Experimental Group (EG), which received therapy with NeuronUP, plus their conventional occupational therapy sessions.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (EG) (Experimental): Experimental Group (EG), which received therapy with NeuronUP, plus their conventional occupational therapy sessions.
  Interventions: Procedure: Conventional occupational therapy sessions + NeuronUP
- Control Group (CG (Active Comparator): Control Group (CG), which received their usual sessions of conventional occupational therapy.
  Interventions: Procedure: Conventional occupational therapy sessions

INTERVENTIONS:
Procedure: Conventional occupational therapy sessions + NeuronUP — Occupational therapy sessions are based on cognitive stimulation, manipulative skill training and psychomotor skills. In addition, 2 sessions per week are conducted with two Nintendo Switch games.
  Arms: Experimental Group (EG)
Procedure: Conventional occupational therapy sessions — Occupational therapy sessions are based on cognitive stimulation, manipulative dexterity training and psychomotor skills.
  Arms: Control Group (CG

SUMMARY:
Introduction: New technologies are a support in the rehabilitation of users. The therapeutic approach to cognitive rehabilitation encompasses a variety of techniques, among which traditional occupational therapy stands out. This modality includes a series of interventions such as cognitive stimulation through the use of cards, functional activities, psychomotor exercises, the application of sensory stimuli and the incorporation of music therapy. An additional alternative is to integrate a cognitive stimulation program such as NeuronUP, which is a computerized tool. This integration can increase adherence to treatment and contribute to preserving or improving the individual's cognitive functioning and improving quality of life.

Objective: The objective established for this study was to verify whether the combination of occupational therapy with the NeuronUP computer program improves or maintains the cognitive status and quality of life of users with Alzheimer's disease. In addition, to determine whether the use of this program leads to greater adherence to treatment by patients.

Material and methods: This is a randomized clinical trial. Participants' cognitive status will be assessed using the MEC (Mini Cognitive Examination) tool, cognitive skills using the LOTCA (Loewenstein Occupational Therapy Cognitive Assessment), and perceived quality of life using the Whoqol-Bref questionnaire. At the end of treatment, the CSQ-8, a tool designed to determine the degree of user satisfaction, will be administered.

ELIGIBILITY:
Inclusion Criteria:

* Adult men or women, aged 65 years or olde.
* Not present severe cognitive impairment, measured through the Mini Cognitive Examination test (MEC>22 points).
* To reside permanently in the Nursing Home.
* Attend Occupational Therapy sessions regularly.
* Have adequate manual dexterity to be able to use a Tablet.
* Agree to participate voluntarily in the study.

Exclusion Criteria:

* Having severe cognitive impairment, as measured by the Mini Cognitive Examination (MEC<22 points).
* Having comorbid diagnoses such as stroke, brain tumours or heart disease, among others.
* Not attending Occupational Therapy sessions regularly.
* Poor adherence to the treatments offered at the centre.
* Not agreeing to participate voluntarily in the study.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 35 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
World Health Organization WHOQOL-BREF | Pre-intervention and post-intervention (up to 1 week)
  Self-administered questionnaire, assesses the general perception of quality of life and general perception of health. It is composed of four domains: physical health, psychological health, social relationships and environment. A higher score on this scale indicates a higher quality of life. Potential scores for all domain scores, therefore, range from 4-20
Mini Cognitive Examination (MEC) | Pre-intervention and post-intervention (up to 1 week)
  This test provides information about a person's cognitive state. By means of the score obtained, cognitive impairment can be perceived, being useful for screening purposes. The scores are: No impairment (between 24 and 35 points); probably moderately impaired (between 23 and 18 points); and severely impaired (less than 18 points).
Loewenstein Occupational Therapy Cognitive Assessment (LOTCA) | Pre-intervention and post-intervention (up to 1 week)
  Tool adapted and validated for the Spanish population that assesses cognitive skills in four areas: orientation, visual and spatial perception, visual motor organisation and thinking operations. Scores range from 1 to 4, with the highest score being the best.

SECONDARY OUTCOMES:
The Client Satisfaction Questionnaire-8, CSQ- | Post-intervention (up to 1 week)
  Self-administered questionnaire used to evaluate satisfaction with the care services received, it consists of 8 questions. Items are scored on a Likert scale from 1 (low satisfaction) to 4 (high satisfaction). Total scores range from 8 to 32, with higher scores indicating greater satisfaction.

CONTACTS AND LOCATIONS:
Locations (1):
- Physiocare Madrid Clinic, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No